

## STUDY PROTOCOL

## with

# STATISTICAL ANALYSIS PLAN

# Prevention and Risk: Treatment with a new emphasis on Relationships (Project Partner)

## NCT03396367

Sponsor: National Institute of Drug Abuse (NIDA)

**Principal Investigator:** Tyrel J. Starks, PhD

Professor

Hunter College

City University of New York

New York, NY

Version Date: January 1, 2024



# **Table of Contents**

| STUDY DESIGN | |
|---|---|
| STUDY TIMELINE | |
| STUDY POPLUATION | |
| Inclusion and Exclusion Criteria: | |
| Contact Information | |
| STUDY PROCEDURES | ε |
| Enrollment Procedures | |
| Informed Consent Process | |
| Post-COVID: Participants review written consent info baseline survey link directs participants to a landing the beginning of the baseline assessment, study staf and confirms age eligibility via Zoom. After reviewing their consent/assent to participate. A copy of the eleparticipant upon request. | page containing detailed consent information. At f provides an oral review of consent information g this information, participants are asked to affirm ectronic consent form is emailed to the |
| Randomization Process/Systems | 8 |
| Schedule of Assessments | <u>S</u> |
| Managing and Tracking Study Visits | 10 |
| Retention and Follow Up | 11 |
| Specimen Collection Pre-COVID | 11 |
| Incentives and Compensation | 12 |
| MEASURES | 17 |
| CASI Measures | 17 |
| INTERVENTION PROCEDURES | 13 |
| Intervention Monitoring | 16 |
| DATA MANAGEMENT AND ANALYSIS PLAN | 17 |
| Data Management and Data Quality | 17 |
| Quantitative Analysis Plan | 19 |
| Moderation/mediation analyses | |
| Qualitative analysis of intervention feedback | |
| Power analyses | 21 |
| Equivalency Checks | 22 |



| IMPLICATIONS AND LIMITATIONS | 22 |
|------------------------------------|----|
| Policy/Methodological Implications | 22 |
| Primary limitations | 22 |
| SAFETY MONITORING PLAN | 23 |
| Adverse Events Reporting | 23 |
| ETHICAL CONSIDERATIONS | 23 |
| Informed Consent Process | 23 |
| REFERENCES | 25 |



#### **STUDY ABSTRACT**

DESIGN: The study utilizes a randomized control trial design, with two

conditions (the experimental PARTNER intervention and an attention-matched Education control) receiving equal

allocation.

SAMPLE SIZE: 240 Sexual minority men (SMM) (18-29) who are in a same

gender relationship. Or 30-34 if they are in a relationship with a

partner who is 18-29

POPULATION: HIV negative SMM who have used drugs in the past 30 days,

and who have engaged in CAS in the past 30 days with a casual partner, a serodiscordant main partner, or a non-monogamous

main partner.

STRATIFICATION: The study will employ a stratified block randomization

procedure with will equate study conditions based upon 1) age discrepancy between partners, 2) relationship length, and 3)

race and ethnicity using Qualtrics.

DATA COLLECTION: Participants have the options to first complete a CASI at home

before their BL appointment (or during BL if they have not done so beforehand). All other aspects of data collection occur at Hunter College. A second CASI survey will also be administered at the BL appointment. Time line follow back interviews to assess drug use, sexual behavior and PrEP adherence (where applicable) will at all assessments. Drug screening and PrEP adherence will be accomplished by obtaining fingernail samples from participants at all assessments. Blood will be collected for

testing PrEP medication adherence. STI testing will be

accomplished by collecting urine and rectal samples at BL, 6m, and 12m. HIV testing will be conducted at BL, 6m, and 12m.

**Post-COVID:** Participants receive a CASI link via email and an athome STI and HIV testing kit, a dried blood spot (DBS) collection kit for PrEP adherence, and a fingernail collection kit for drug screening (via regular mail) prior to assessment appointments.



All other aspects of data collection occur remotely via HIPAA-compliant Zoom.

**OBJECTIVES:** 

- 1) Evaluate the efficacy of PARTNER in regards to three primary outcomes: 1) PrEP uptake and adherence 2) sexual transmission risk behavior and 3) drug use.
- 2) Identify individual and relationship factors which moderate/mediate intervention efforts.
- 3) Gather ideographic data to inform a future effectivenessimplementation study.
- 4) Validate the use of fingernail assays as a biological marker for PrEP adherence.



#### STUDY DESIGN



Figure 3. Participation timeline

- <sup>a</sup> To detect drug use for all participants and PrEP adherence for those on PrEP.
- <sup>b</sup> Gathered only for those on PrEP

#### **STUDY TIMELINE**





#### STUDY POPLUATION

#### Inclusion and Exclusion Criteria:

Participants who express interest in PARTNER must demonstrate the following inclusion criteria to be enrolled in the study:

- 18 29 years old; or 30-34 with a partner who is 18-29 (inclusive)
- Have a main partner who is another male for 1 month or longer
  - Main partner must be 18 years old or older
- Be HIV negative (as confirmed by rapid test)
- Have used drugs in the past 30 days
- Have engaged in TRB in the past 30 days
  - Defined as CAS with a casual partner and/or CAS with a non-monogamous or serodiscordant main partner
- Live in the NYC metropolitan area (Enrollment expanded nationwide in the US in September 2022.)
- Speak English

Participants are excluded from the study if they any indicate the following:

- Any signs of serious mental illness or cognitive deficit
- History of intimate partner violence with their main partner or feel unsafe in their current relationship.

#### **Recruitment and Screening**

We utilize a multi-faceted recruitment effort including both active and passive approaches. Our previous research focused on MSM in relationships has indicated that online recruitment is particularly effective at reaching this target population. We anticipate enrolling 6 new participants each month. Contacts obtained through our online screener will be contacted for scheduling. Contacts that come from the online master screener will be sent 2 emails with links to take our study specific screener. Once scheduled, participants are sent their at-home survey link. They do not have to complete this survey beforehand, but we do remind them two times before their baseline appointment to complete it as it cuts down on the time they need to be in the office.

**Post COVID:** Contacts obtained through our cross project online screener are contacted to schedule a baseline appointment on Zoom. Before the baseline appointment, the study staff contacts the participants via text or phone call to obtain preferred mailing address for testing kit shipments, confirm contact information, and obtain participant PrEP status in order to ship the correct laboratory testing kit. The baseline assessment is scheduled and study staff sends participants their at-home survey link and orders their STI/HIV testing kits. Participants must



complete this survey and have received their testing kits before their remote baseline appointment can occur.

#### **Contact Information**

Once they are screened eligible through our online screener, participants' contact information is collected and they are asked if messages can be left at the numbers provided or if text can be sent. Study staff do not leave messages or send text messages unless expressly permitted to do so by the participant, which is documented on the participant Locator Form and Access DB.

#### STUDY PROCEDURES

## **Enrollment Procedures**

Participants are considered enrolled in the study when they have completed informed consent. Randomization occurs immediately after the baseline appointment.

#### **Informed Consent Process**

Details of the study are reviewed with the prospective study participant by a research assistant who is trained and cleared to conduct assessments and is knowledgeable about the research study. This discussion is a critical component of the consent process and the prospective study participant will be given adequate time for this discussion and to read the written consent form. The research assistant is available to answer questions about the study including participant responsibilities, benefits, risks, and alternatives. The participant reviews the consent form and it is signed and dated by both the participant and study staff member conducting the assessment. A copy of the signed consent form will be given to the participant and the original will be kept securely by the project coordinator separate from other assessment materials.

<u>Post-COVID:</u> Participants review written consent information prior to their baseline appointment. The baseline survey link directs participants to a landing page containing detailed consent information. At the beginning of the baseline assessment, study staff provides an oral review of consent information and confirms age eligibility via Zoom. After reviewing this information, participants are asked to affirm their consent/assent to participate. A copy of the electronic consent form is emailed to the participant upon request.

## **Randomization Process/Systems**

Participants are randomized at the end of their baseline assessment into one of two intervention conditions: 1) delivery of the 4 session PARTNER intervention or 2)



delivery of 4 education sessions. Each participant's condition is tracked in the access tracking database maintained by the project manager.

The study employs a stratified block randomization procedure with equate study conditions based upon 1) age discrepancy between partners, 2) relationship length, and 3) race and ethnicity using Qualtrics.

#### Schedule of Assessments

Sessions occurs approximately <u>once per week</u> for three weeks beginning one week after completion of the baseline assessment and session 1. There is a 12 week window for intervention completion, i.e. all four sessions must be completed within 12 weeks of the baseline assessment.

Participants complete the first follow-up assessment 3 months after the baseline, and subsequent follow ups at 6, and 9 months after baseline with a final appointment scheduled for 12 months following the baseline appointment. Study staff should aim to schedule and complete these follow-ups as close as possible to each target date. To keep track of longitudinal data collection dates, assessment visit windows will be defined as 15 days prior and after the target as "in window." The assessment visit window for the 12 month follow-up ends 30 days after the target date. Site study staff should prioritize the completion of sessions before the first follow-up assessment, and should not schedule this follow-up less than 12 weeks after baseline if a participant is available to complete any additional sessions first.

**Post-COVID:** The 12-month assessment window ends 60 days after the target date.

| Component | Baseline | Session 1 | Session 2 | Session 3 | Session 4 | 3-Month<br>Follow-Up | 6-Month<br>Follow-Up | 9-Month<br>Follow-Up | 12-Month<br>Follow-Up |
|---|---|---|---|---|---|---|---|---|---|
| Informed Consent | Х | | | | | | | | Х |
| Randomization | Х | | | | | | | | |
| CASI | Х | | | | | Х | Х | Х | Х |
| TLFB | Х | | | | | Х | Х | Х | Х |
| HIV Testing (Rapid for those not on PrEP – | Х | | | | | | Х | | Х |



| Architect for those on PrEP) | | | | | | | |
|---|---|---|---|---|---|---|---|
| STI Testing | Х | | | | Х | | Х |
| Fingernail Assay for Drugs | Х | | | Х | Х | х | Х |
| Dried Blood Spot<br>(For those on PrEP) | х | | | Х | Х | Х | Х |
| PrEP Video | | X | | | | | |
| Video Recall Survey for those who seen the Video | | | Х | х | | | х |
| Session feedback | | | Х | | | | |
| Qualitative Interview | | | | | | | х |

## **Managing and Tracking Study Visits**

There are two different types of visits during the study timeline:

Session Visits: Session visits refer to both the four education and four intervention sessions. Intervention sessions are conducted by trained and cleared MI-trained clinicians. Intervention sessions will be managed by the clinicians with their individual study participants. Clinicians will notify site study staff of whether visits were completed for tracking purposes, provide receipts for session compensation to site study staff, and upload audio files to Project Partners respective folder on the M drive as per study procedures. Education sessions are conducted by trained and cleared health educators. Education sessions will be managed by the educators with their individual study participants. Educators will notify site study staff of whether visits were completed for tracking purposes, provide receipts for session compensation to site study staff, and upload audio files to Project Partners respective folder on the M drive as per study procedures.

**Research Visits:** Research visits include all assessments including the baseline visit, the post-test assessment, and all other follow-up assessments. All participants, in either condition, are expected to complete <u>five</u> assessment visits as part of full participation in the study.

Study staff will schedule participants during times that they will be available or will contact other staff to ensure coverage for appointments. Study staff will also ensure that there is available space to conduct these assessments.

Future visits should be scheduled during the study visit. Study staff are expected to keep in touch with participants and remind them of the upcoming visit or reschedule if



needed. A reminder call should be made the day before a participant is due to come in for their visit (or the Friday before a Monday visit).

#### **Retention and Follow Up**

**Session visits:** For participants who are actively taking part in the PARTNER intervention or the Education control condition, site study staff will not add an additional level of outreach to the procedures.

## **Specimen Collection Pre-COVID**

HIV testing will be performed at the baseline using the HIV 4<sup>th</sup> Generation assays and those will be administered following the below criteria:

- 1- Participants on PrEP, upon PrEP self-report confirmation will provide 1 tube of blood to send to the LAB for HIV Confirmatory testing with Architect equipment to avoid any inaccurate test results as a result of PrEP drugs in blood. Results are downloaded from the LAB's web portal.
- 2- Participants NOT on PrEP, will be administered a rapid HIV Test named "Determine Ab/Ag" which detects HIV antibodies and antigen P24 (the last one is a very sensitive part of this specific test and can detect early acute HIV infections).

At baseline we test for Urethral and Rectal Gonorrhea & Chlamydia presence. The testing method for Urethral G&C will involve the participant urinating in a sterile urine collection cup then to pipette just a portion of that urine sample into a sample tube in order to be sent for testing to Sunrise medical Laboratory. For Rectal detection we will provide the participant with an anal swab collection kit, and send the specimen for STI detection to Sunrise Medical Laboratory.

We will collect participant's fingernails and potentially toenails in case the sample is not enough, to test illicit drug use in the last 6 months, this 5-Panel drug assay will be conducted by USDTL Laboratory.

A second vial of blood will also be collected at the same time as the HIV test vial with participants reporting being on PrEP, to perform dried blood spot (DBS) cards to test for PrEP adherence, which will be sent to Colorado Antiviral Pharmacology Laboratory.

## **Post-COVID Specimen Collection**

HIV and STI tests are completed using tests shipped and processed by Molecular Testing Labs (MTL). Prior to the RA administered portion of the baseline assessment and 6- and 12-month follow-ups, participants are mailed a package containing an athome OraQuick testing kit for HIV, self-administered rectal and urethral gonorrhea and chlamydia testing kits, one dried blood spot (DBS) card (if on PrEP), collection



materials (alcohol prep pads, lancets, gauze pad, and adhesive bandages), an instruction card, and a postage-paid shipping envelope. During the RA administered portion of the baseline, 6M, and 12M, the RA will review instructions and demonstrate the collection procedure. The RA will then remain on the Zoom call to provide any additional guidance as needed during the collection procedure. Participants will then place the collected specimens in the addressed envelope for shipping to the lab for processing. Participants will also be mailed a fingernail collection kit to examine drug use rates during all assessments.

## **Incentives and Compensation**

Participants will be compensated up to \$380 for full participation in the study. They will receive:

\$50 for completing a Baseline assessment.

\$20 for each completed session (up to \$80 total).

\$60 for completing a 3-Month Follow-Up Assessment.

\$60 for completing a 6-Month Follow-Up Assessment.

\$60 for completing a 9-Month Follow-Up Assessment.

\$70 for completing a 12-Month Follow-Up Assessment. (**Post-COVID**: \$100 for completing a 12-Month Follow-Up Assessment)



#### INTERVENTION PROCEDURES

The PARTNER intervention comprises 4 sessions of Motivational interviewing (MI) to address 3 target behaviors that correspond to the study's primary outcomes: drug use, PrEP uptake/adherence, and HIV transmission risk. Miller and Rollnick suggested that 4 processes are ongoing during an MI session: engagement (establishment of a therapeutic alliance), focusing (clarification of session goals), evoking (eliciting speech in favor or change while softening arguments for the status quo), and planning (the identification of action steps that can be taken toward the accomplishment of an identified goal). The salience of these various processes is dependent upon the duration of the relationship between the interventionist and the participant as well as the client's stage of change.

The first session emphasizes the engaging process. It begins with an introduction to the participant followed by an exploration of participant's primary relationship, understanding how he and his partner handle sex outside their relationship, and enhancing motivation to reduce both drug use and HIV infection risk. This conversation then focuses on what strategies, if any, the participant and his partner use to manage their HIV risk. The interventionist then seeks to evoke motivation to reduce HIV related risk, potentially through PrEP uptake or adherence. The values card sort activity is utilized midway through the session to integrate a conversation about how the participant's values are expressed in his relationship and the decisions made around HIV prevention. The second session engages the participant in a review of the previous week and then transitions to focus on drug use. The interventionist seeks to evoke motivation to reduce drug use, with particular attention given to how the participant's relationship partner feels about use. The third session integrates a focus on the links between drugs and CAS with main and casual partners, PrEP, and presents video-based modeling to enhance communication skills. This facilitates a longer discussion about planning toward any identified goals. The interventionist gives particular attention to the role of relationship partners during the planning phase. The final session engages the participant in a review of the previous week. The session then proceeds to review the participant's perception of the overall intervention process with emphasis on successes and challenges. The session emphasizes the planning process by inviting the participant to identify long-term goals related to the target behavior and develop plans to accomplish these goals. A discussion of relevant resources and referrals occurs during this time.



PARTNER incorporates a video-based approach to relationship skill building with a structured series of debriefing questions asked by the MI provider after the video is viewed. The video utilized was comprised of 3 scenes, each depicting a different couple. It is integrated into Session 3 of the intervention and serves a dual purpose. First, it provides information specific to PrEP. Each scene depicts either a nonmonogamous or serodiscordant couple discussing PrEP and HIV prevention. In this way, participants viewing the video see men in relationships with men talking about reasons why PrEP might be relevant, while also receiving basic information about PrEP and its efficacy. Second, the videos directly teach communication skills through modeling. Each scene is divided into 2 parts. In the initial portion of the scene, the couple makes a specific communication error. Midway through the scene, a narrator interrupts the couple, explains their error, and suggests an alternative strategy. The scene then continues, and the couple communicates more effectively.

## **SESSION 1: Focus on CAS with main and casual partners**

- Opening statement provide information as appropriate; set the stage for collaboration; introduce target behaviors
- Values Card Sort Use Open Questions and Reflections, close with a major Summary
- Use strategies for eliciting change talk & managing discord
- At the end of the session, offer a closing summary highlighting any change talk or steps towards change; evoke commitment to attend future session

#### **SESSION 2: Focus on drug use**

- Opening statement highlight any change talk or plan from previous session; introduce second target behavior and collaborate on setting session agenda with client
- Briefly revisit last session's topic and check for any changes or recent events since you last met
- Ask permission to discuss second target behavior
- Use strategies for eliciting change talk and managing discord
- Offer to help in creating a strategy to change target behavior
- Offer a closing summary at the end of the session, highlighting change talk and any steps taken towards change



## SESSION 3: Focus on drugs, CAS with main and casual partners, and PrEP

- Opening statement: Highlight and integrate change talk on both target behaviors and any ideas or goals the client has articulated around these behaviors; work collaboratively to set the agenda for the session
- Ask the client where they would like to go from here; or, ask permission to discuss collaborating on a change plan together
- Evoke client's ideas about change; build on past success; evoke and reinforce selfefficacy for taking steps towards change
- If appropriate, use the Ask-ask-tell-ask-reflect approach for offering information or suggestions; if offering suggestions be sure to reinforce client autonomy and offer a menu of options
- Collaborate with the client to build a change plan that reflects their goals, priorities and readiness to change; elicit the client's ideas about how the plan could be carried out, when the steps will occur and why these changes are important
- Offer a closing summary highlighting change talk and briefly reiterating the basic plan; reinforce client autonomy; remind the client that the next session will be focused on moving ahead independently.

## SESSION 4: Focus on drugs, and CAS with main and casual partners

- Opening Statement: Summarize the plan developed previously and collaborate on setting the session agenda; introduce termination / last YMHP session;
- Check in on how the plan has been going since you last met; use strategies for evoking change talk / managing discord as appropriate; affirm client for any steps towards change;
- Evoke client's ideas about how to improve or adapt the plan; evoke and reinforce commitment for maintaining the plan moving forward
- Evoke client's ideas about what to do should problems arise in the future; develop a 'backup plan' as appropriate
- Summarize progress over the 4 sessions and termination

**Post-COVID:** The PARTNER intervention is administered via Zoom following the procedures outline above. Interventionists share their screen with participants when needed to present video components of the intervention. The values card sort activity is completed using a version of the task programmed into Qualtrics. Interventionists share their screen, and participants direct them how to sort values.



## **Education Intervention (Control Condition)**

The education intervention is administered one-on-one by a health educator. The sessions are guided by a PowerPoint presentation that helps to insure fidelity of delivery while also increasing the participant's engagement through the integration of pictures, animation, and video. The presentation is viewed on a personal computer located in the intervention room. Dual monitors are used to ensure that both the educator and participant can readily view material.

The condition comprises of 4 sessions of health education addressing sexual risk and drug use. The sessions utilize a mixture of modalities including lecture, question and answer, and video. Session 1 focuses on HIV risk and prevention. Lecture content is supplemented by videos focusing on HIV transmission generally and HIV prevention strategies among gay and bisexual men specifically. Session 2 is focused on drug use. Information about the biological effects of drug use is largely provided through videos. Lecture content and discussion questions focus on the impact of drug use within the local gay community. Session 3 examines the intersection of drugs and sex in the local gay community. Education content also focuses on mitigating the risks associated with having sex while intoxicated. Session 4 again focuses on drug use with video and lecture-delivered content describing the signs and warnings of potential substance use disorders.

**Post-COVID:** The education intervention is administered via Zoom following the procedures outlined above. Health educators share their screen with participants to present PowerPoint slides and review session content.

#### Intervention Monitoring

All sessions will be audio recorded. MI fidelity in the PARTNER intervention will be evaluated using the Motivational Treatment Integrity coding system<sup>141</sup>. We will randomly select 25% of session to be coded. A team of trained coders is maintained and utilized in all NIH-funded studies involving MI-based interventions. The educators for the control condition will undergo similar fidelity procedures in which 25% of their education sessions will be evaluated for fidelity. These recordings will be reviewed and matched to a fidelity checklist that outlines the content of the Education session. Successful Education sessions will have accurately discussed at least 90% of the content.



#### DATA MANAGEMENT AND ANALYSIS PLAN

## **Data Management and Data Quality**

Qualtrics, a secure online survey platform which can be accessed from computers on site, is used to administer survey measures during in-person appointments. Qualtrics is sufficiently flexible to permit the use of a wide range of question and response types.

Qualitative interviews will be recorded, transcribed, and de-identified.

## **MEASURES**

## **CASI Measures**

| | Construct | Measure |
|---|---|---|
| Screening | Demographics | NHBS demographics inventory <sup>107</sup> |
| information | Sexual HIV transmission risk | Self-Reported Sexual Behavior |
| | PrEP uptake and related attitudes | PrEP uptake questionnaire <sup>15,68</sup> |
| | Problematic drug use | Drug Abuse Screening Test – 10 <sup>108</sup> |
| | Alcohol and Drug Use<br>Behavior | NHBS Substance Use History<br>Inventory <sup>107</sup> |
| | Partner health behavior | Partner health behavior survey |
| IMB factors | Knowledge: Drug use | Drug use knowledge questionnaire |
| | Knowledge: HIV infection (including condom and PrEP supplement) | Brief HIV knowledge questionnaire 109 |
| | Motivation: Drug use | Decisional Balance - Club Drugs <sup>110</sup> |
| | Motivation: Condom use | Decisional Balance - Unsafe Sex <sup>110</sup> |
| | Motivation: PrEP | Decisional Balance - PrEP |
| | Behavioral Skill: Drug use | Drug Taking Confidence<br>Questionnaire <sup>111</sup> |
| | Behavioral Skill: Condom<br>use | Condom use self-efficacy scale <sup>112</sup> |
| | Behavioral Skill: PrEP | Adapted Adherence Self-Efficacy Scale <sup>1</sup> |
| Individual | Condom attitudes/beliefs | Adapted condom attitudes scale <sup>32</sup> |
| functioning | Anxiety and Depression | Brief Symptom Inventory <sup>114</sup> (subscales) |
| | Experiences of stigma | Everyday discrimination <sup>115</sup> |
| | Intimate Partner Violence (IPV) | IPV among gay and bisexual men 116 |
| | Problematic alcohol use | Alcohol Use Disorders Identification Tes<br>(AUDIT) <sup>117</sup> |
| | Self-reported STI and HIV | |
| | - | |



| | testing history; PrEP; and ART | |
|---|---|---|
| Relationship functioning | Relationship satisfaction, cohesion, consensus & affectional expression | Dyadic adjustment scale <sup>118</sup> |
| | Interpersonal | Interpersonal Communication |
| | Communication Skills | Competence Scale <sup>119</sup> |
| | Partner communication strategies | Communication patterns questionnaire <sup>120</sup> |
| | G | Sexual communication <sup>121</sup> |
| | Couples HIV Coping | Perceived severity of HIV infection <sup>122</sup> Preferences for sexual health outcomes <sup>122</sup> |
| | | Couple efficacy to reduce HIV threat 122 |
| | Stigma directed at the relationship | Relationship marginalization <sup>123</sup> |
| | Relationship Control & Dominance | Sexual Relationship Power Scale (SRPS) <sup>124</sup> |
| | Attitudes about Sexual<br>Agreements | Sexual Agreement Investment Scale (SAIS) <sup>100</sup> |

#### **Primary outcomes**

**Drug use.** During TLFB interviews, participants indicated whether they used any of 10 different drug types. Responses produced two count variables indicating the number of days participants used cannabis and the number of days they reported the use of any illicit drugs, including: cocaine, crack, methamphetamine, ecstasy, ketamine, GHB, and psychedelics. Self-reported drug use was corroborated by fingernail assay. See supplemental material for details.

**Current PrEP uptake** was assessed using a single survey item, "Have you ever been prescribed PrEP (HIV pre-exposure prophylaxis)?" Participants taking PrEP reported days they missed their PrEP on the TLFB interview. Responses were used to create a dichotomous variable indicating whether or not participants took PrEP on at least 57% of days (corresponding to at least 4 days out of 7 on average). Self-reported PrEP adherence was corroborated with DBS results. See supplemental material for details.

**Sexual HIV TRB.** During TLFB interviews, participants indicated days they had (insertive or receptive) anal sex with any casual partners and whether a condom was used. Responses were aggregated to create a variable indicating the number of times the participant had CAS with a casual partner. If participants were prescribed PrEP and reported missing 13 doses or fewer, they were assigned a value of 0, reflecting that the use of PrEP on at least 4 of 7 days is sufficient to achieve reductions in HIV TRB (28). Self-reported CAS with casual partners was corroborated by bacterial STI diagnosis. See supplemental material for details.



#### **Putative moderators**

**Relationship satisfaction** was assessed using the approximation to ideal subscale of Kurdek's (29, 30) Multiple Determinants of Relationship Commitment Inventory (MDRCI). The subscale consists of 4 items (e.g., "My current relationship comes close to matching what I would consider to be my ideal relationship"). Response options ranged from 1 (strongly disagree) to 5 (strongly agree). Total score reliability was good (Cronbach's  $\alpha = .848$ ).

**Communication skills.** Self-disclosure, social anxiety, assertiveness, and empathy subscales of the Interpersonal Communication Competence Scale (31) assessed aspects of communication skills. Each subscale was assessed by 3 statements (e.g., "I can put myself in others' shoes" and "It's difficult to find the right words to express myself"). Participants evaluated each statement using a 5-point scale Likert-type scale ranging from 0 ("Almost never") to 4 ("Almost always"). Total score reliability was good (Cronbach's  $\alpha = .787$ ).

## **Quantitative Analysis Plan**

The primary hypotheses are that SMM receiving the PARTNER intervention will be more likely to initiate and/or be adherent to PrEP throughout the follow up period. As a result, it is hypothesized they will have a lower probability of TRB. In addition, it is hypothesized that the PARTNER intervention will be associated with lower levels of drug use (number of use instances) compared to the education condition.

## **Corroboration of self-reported behavior with biomarkers**

Self-reported drug use was corroborated by fingernail assays. At baseline and all follow-ups, at least 80% of participants who tested positive for cannabis indicated at least one instance of cannabis use. In addition, at least 60% of those who did not test positive for cannabis on fingernail assays indicated they used cannabis at least once. At baseline, and all follow-ups, at least 55% of those who tested nail positive for cocaine, crack, or amphetamine use reported at least one instance of illicit drug use. In addition, 12% of those who did not test positive for illicit drug use on nail samples self-reported the use of at least one drug.

Self-reported PrEP adherence was corroborated with DBS results. At baseline and all follow-up time points, no fewer than 69% of participants who reported taking their PrEP on 57% of days or more had a DBS test result of 700 units of TFV-DP per DBS punch or greater at all follow-up time points. One participant at baseline and another at the 3month follow-up reported missing more than 57% of their PrEP but produced a DBS result of 700 units of TFV-DP per DBS punch or more.

Self-reported CAS with casual partners was corroborated by bacterial STI diagnosis. Participants were indicated as having a bacterial STI if they received a positive result for rectal or urethral gonorrhea or chlamydia at baseline, 6, or 12-month follow-up or if they self-reported receiving a diagnosis in the past 3 months at any assessment point. At baseline, 30.5% of those who



reported CAS with a casual partner had a bacterial STI compared to 7.7% of those who did not. Similarly, 44.2% of participants who reported having CAS with a casual partner at either the 3 or 6-month follow-up had a bacterial STI, compared to 23.9% of those who did not. Finally, 39% of those who reported having CAS with a casual partner at the 9 or 12-month follow-up had a bacterial STI compared to 9.5% of those who did not.

## **Detailed analytic plan**

A series of bivariate analyses ( $\chi 2$  tests of independence and independent samples t-tests) conducted in SPSS (version 29) evaluated the success of randomization and the presence of differential attrition. The generalized linear model function in SPSS was used to evaluate between-condition differences in baseline frequency of primary outcomes with count distributions (cannabis use days, other illicit drug use days, sexual HIV TRB) and baseline odds of PrEP uptake (a dichotomous variable).

Outcome analyses were conducted using piece-wise latent growth curve (LGC) models following procedures outlined by Chou et al. Growth trajectories over time following the delivery of an intervention may be characterized by a large initial response followed by a more sustained trajectory with a less dramatic slope. Piece-wise LGC models quantify this kind of trajectory using two slopes. Slope 1 quantifies the change from baseline to the immediate post-test (3-month follow-up). Meanwhile, Slope 2 quantifies the trajectory over the post-intervention follow-up period.

Two models were calculated for each outcome. Model 1 included the main effect of treatment on growth factors. Model 2 added the main effects of moderators (communication skills and relationship quality) as well as the interaction terms between these moderators and the main effect of treatment.

Several considerations led to the inclusion of model covariates. Consistent with guidance for the analysis of data from randomized controlled trials that utilize stratified randomization (16), stratification variables were included as covariates in regressions predicting latent growth factors. The COVID-19 pandemic and recovery corresponded with changes in substance use and sexual behavior among SMM. To account for this, models incorporated a dichotomous, timevarying predictor indicating whether an assessment occurred before or after March 2020. All models were calculated using full-information maximum likelihood estimation in Mplus Version 8.0. This permitted the retention of all randomized cases consistent with the intent-to-treat paradigm. Model significance was evaluated using a robust log-likelihood  $\chi 2$  test comparing the log-likelihood of the specified model to a null-model – in which all structural coefficients associated with the regression of latent growth factors on condition and site were constrained to be zero. Where model results were significant, the effect of the PARTNER intervention was evaluated by examination of regression parameters for Slopes 1 and 2. Given the directional nature of hypotheses, single-sided p-values were used to determine the



significance of the intervention effect. When evaluating the significance of putative moderators and associated interaction terms, two-sided p-values were used.

## **Power** analyses

We utilized the *Test for the Ratio of Two Negative Binomial Rates* module in PASS 19 to evaluate power to detect between-condition differences in drug use frequency at any one follow-up time point. Power (1-beta) was set to .80 and the probability of type II error (alpha) was set to .05. The number of exposures was set to 30 (the number of days of use assessed in the TLFB). The rate of use in the education condition was set to 3, 6, and 9. Meanwhile dispersion values of 1, 2, and 4 were tested. Power was highest at low levels of dispersion and high based rates of use in the education condition. Under these circumstances, the study has power=.80 to detect a rate ratio of 0.70 or a 30% reduction in drug use instances. At high levels of dispersion and low base rates, the study would be expected to detect a rate ratio of 0.48.

Power to detect differences in HIV transmission risk behavior was calculated in 2 ways. First, using procedures similar to those described for drug use, the study has power to detect a rate ratio between 0.48 and 0.69 in the number of CAS events in the absence of PrEP. This calculation tested average rates of CAS in the absence of PrEP in the education condition of 1, 3, and 5 instances and dispersion was tested at values of 1, 2, and 4. Power to detect significant differences in the odds of a positive STI test was calculated using the *inequality tests for 2 proportions in a repeated measures design* module [60]. Analyses specified 4 waves of data, power (1-beta) was set to .80, and the probability of type II error (alpha) was set to .05. Autocorrelation (rho) was permitted to vary between .25 and .75. The proportion of positive STI diagnosis in the education condition was tested at values of .13, .10, and .07. Power declined as rho increased. Power increased with the proportion of positive diagnoses in the education condition. Analyses suggested that the study is adequately powered to detect large effects, associated with an odds ratio between 0.20 (under the least favorable conditions) and 0.32 (under the most favorable).

Power to detect differences in PrEP uptake was similarly calculated using the *inequality tests for 2* proportions in a repeated measures design module [60]. Analyses specified 4 waves of data, power (1-beta) was set to .80, and the probability of type II error (alpha) was set to .05. Autocorrelation (rho) was permitted to vary between .25 and .75. We estimated that on average 35% of the education condition would be on PrEP during the follow-up period. The proposed sample is sufficient to detect an odds ratio



of 1.90 even at the highest values of rho, which corresponds to approximately 51% of the PARTNER condition initiating PrEP. With regard to adherence, assuming approximately 100 participants (45% of the sample assuming 80% retention) are on PrEP at any follow-up point and 75% of the control condition is adherent to their PrEP medication (Cronbach alpha=.05; and  $\rho$ =.25 to .50), results suggested that the study has power=.80 to detect an odds ratio of approximately 3.0.

## **Equivalency Checks**

We will strive to ensure that randomization will not produce any significant differences in participant characteristics that require control in subsequent longitudinal analyses. Baseline cross-site variance in participant characteristics will be assessed using standard tests of mean differences for both biological markers and self-reported measures of substance use, TRB, and PrEP uptake/adherence. Assignment differences in baseline demographics will be assessed using standard non-parametric measures of association. Any observed differences will be controlled for in subsequent models.

#### IMPLICATIONS AND LIMITATIONS

## **Policy/Methodological Implications**

This application has focused implications for the\_biomedical prevention of HIV in a highly vulnerable population as well as broad methodological implications for PrEP research. The proposed project tests an intervention which addresses PrEP uptake in a high-priority population for whom no existing interventions are tailored (partnered SMM meeting CDC criteria for PrEP candidacy). It therefore addresses PrEP uptake and adherence (critical steps in the cascade) for an under-served and highly vulnerable population. Furthermore, the secondary aims of this proposal include the validation of fingernail assays to assess PrEP adherence. This innovation has broad implications for the study of PrEP.

## **Primary limitations**

1) The absence of data from relationship partners. The use of individual (rather than dyadic) intervention is intended to enhance scalability. Participants will report relationship functioning as well as their perception of their partners' drug use, sexual behavior, PrEP uptake (see APPENDIX B; Partner health behavior survey). This will provide proxy data which can inform future studies. 2) Limited data on the efficacy of the PARTNER intervention. We have completed all aspects of intervention development and established the acceptability/feasibility of PARTNER. The need for pilot efficacy data is reduced by the fact that PARTNER incorporates all aspects of YMHP, which has demonstrated efficacy<sup>16</sup>, and the use of a control condition which has been employed in previous NIH funded trials<sup>16</sup>. 3) Recruiting partnered SMM. A strong infrastructure exists to support recruitment efforts. We have developed recruitment



protocols and tracking systems that have facilitated a detailed examination of the efficiency of recruitment efforts<sup>18,105,106,146</sup>. We have also specifically examined issues related to dyadic vs. individual participation in research on partnered MSM<sup>18</sup>.

## **SAFETY MONITORING PLAN**

## **Adverse Events Reporting**

The Site PI is responsible for the detection and documentation of events meeting the criteria and definition of an AE or SAE. Study staff may ask PI questions concerning adverse events, but must formally report them via email. Information on unexpected events including serious adverse effects (SAEs) will be reported as per the policy of the IRB.

Information to be collected includes the nature, date of onset, stop date, intensity, duration, treatment, causality, and outcome of the event. Pls should follow usual clinical practices for reporting serious, unexpected events related to standard of care. SAEs that occur after 30 days after completion of the study will be collected only if they are considered by the PI to be related to study participation. In addition, any AE resulting in potential participant withdrawal must been reported to the PI prior to participant withdrawal when possible.

PIs must report any Adverse Event to the IRB within five business days of learning of it.

#### **ETHICAL CONSIDERATIONS**

#### **Informed Consent Process**

Site PIs must ensure that participants are fully informed about the purpose, responsibilities of participating and potential risks or other critical issues related to participation in the study. Written informed consent is obtained from every participant or, in those situations where consent cannot be given by participants, their legally acceptable representative, prior to clinical study participation.

The rights, safety, and well-being of study participants are the most important considerations and should prevail over interests of science and society. If there is any question that the prospective participant will not reliably comply with study procedures and/or follow-up, they should not be enrolled in the study.





## **REFERENCES**

- CDC. Preexposure prophylaxis for the prevention of HIV infectionin the United States 2014. A clinical practice guideline. 2014. http://www.cdc.gov/hiv/pdf/prepguidelines2014.pdf. Accessed 4/25/2016.
- 2. Prevention CfDCa. HIV Surveillance Report. In: Prevention CfDCa, ed. Vol 272015.
- 3. CDC. HIV and substance use in the United States. 2013.
- 4. Sullivan PS, Salazar L, Buchbinder S, Sanchez TH. Estimating the proportion of HIV transmissions from main sex partners among men who have sex with men in five US cities. *AIDS*. 2009;23(9):1153-1162.
- 5. Parsons JT, Lelutiu-Weinberger C, Botsko M, Golub SA. Predictors of day-level sexual risk for young gay and bisexual men. *AIDS Behav.* 2013;17(4):1465-1477.
- 6. Salomon EA, Mimiaga MJ, Husnik MJ, et al. Depressive Symptoms, Utilization of Mental Health Care, Substance Use and Sexual Risk Among Young Men Who have Sex with Men in EXPLORE: Implications for Age-Specific Interventions. *AIDS Behavior*. 2009;13(4):811–821.
- 7. Austin EW, Bozick R. Sexual orientation, partnership formation, and substance use in the transition to adulthood. *Journal of Youth and Adolescence*. 2011;41:167-178.
- 8. Marshal MP, Friedman MS, Stall R, Thompson AL. Individual trajectories of substance use in lesbian, gay and bisexual youth and heterosexual youth. *Addiction*. 2009;104(6):974-981.
- 9. Parsons JT, Starks TJ. Drug use and sexual arrangements among gay couples: frequency, interdependence and associations with sexual risk. *Archives of Sexual Behavior*. 2014;43(1):89-98.
- 10. Parsons JT, Starks TJ, Dubois S, Grov C, Golub SA. Alternatives to monogamy among gay male couples in a community survey: implications for mental health and sexual risk. *Archives of Sexual Behavior*. 2013;42(2):303-312.
- 11. Starks T, Millar B, Parsons J. Predictors of condom use with main and casual partners among HIV-positive men over 50. *Health Psychol.* 2015;34(11):1116-1122.
- 12. Hoff CC, Beougher SC. Sexual agreements among gay male couples. *Archives of Sexual Behavior*. 2010;39:774-787.
- 13. Mimiaga MJ, Closson EF, Kothary V, Mitty JA. Sexual partnerships and considerations for HIV antiretroviral pre-exposure prophylaxis utilization among high-risk substance using men who have sex with men. *Archives of Sexual Behavior*. 2014;43(1):99-106.
- 14. Starks TJ. Tailoring and framing biomedical prevention for gay men in relationships. PRIDE 20th Anniversary symposium. HIV research that informs policy: Past, present and future; 2016; New York City, NY.
- 15. John SA, Starks TJ, Rendina HJ, Grov C, Parsons JT. Should I convince my partner to go on Pre-Exposure Prophylaxis? The role of personal and relationship factors on PrEP-related social control among gay and bisexual men. in production.



- 16. Parsons JT, Lelutiu-Weinberger C, Botsko M, Golub SA. A randomized controlled trial utilizing motivational interviewing to reduce HIV risk and drug use in young gay and bisexual men. *Journal of Consulting and Clinical Psychology*. 2014;82(1):9-18.
- 17. Stephenson R, Grabbe KL, Sidibe T, McWilliams A, Sullivan PS. Technical assistance needs for successful implementation fo couples HIV testing and counseling (CHTC) intervention for male couples at US HIV testing sites. *AIDS Behav.* 2016;20:841-847.
- 18. Starks TJ, Millar B, Parsons JT. Correlates of individual versus joint participation in online survey research with same-sex male couples. *AIDS Behav.* 2015;19:963-969.
- 19. Yucel D, Gassanov M. Exploring actor and partner correlates of sexual satisfaction among married couples. *Social Science Research*. 2010;39(5):725-738.
- 20. Cappelle D, Yegles M, Neels H, et al. Nail analysis for the detection fo drugs of abuse and pharmaceuticals: A review. *Forensic Toxicology*. 2015;33(1):12-36.
- 21. Fisher JD, Fisher WA. Changing AIDS-risk behavior. *Psychological Bulletin*. 1992;111(3):455-474.
- 22. Rusbult CE, Van Lange PA. Interdependence, interaction, and relationships. *Annual Review of Psychology.* 2003;54:351 375.
- 23. Rendina HJ, Moody RL, Ventuneac A, Grov C, Parsons JT. Aggregate and event-level associations of substance use and sexual behavior among gay and bisexual men: Comparing retrospective and prospective data. *Drug and Alchol Dependence*. 2015;154:199-207.
- 24. Yu G, Wall MM, Chiasson MA, Hirshfield S. Complex drug use patterns and associated HIV transmission risk behaviors in an internet sample of U.S. men who have sex with men. *Archives of Sexual Behavior*. 2014;44:421-428.
- 25. CDC. HIV Surveillance Report. Vol 242014.
- 26. Centers for Disease Control and Prevention. HIV surveillance report, 2014. 2015;26. http://www.cdc.gov/hiv/library/reports/surveillance/. Accessed December, 2015.
- 27. Erikson EH. *Identity and the life cycle*. New York: Norton; 1980.
- 28. Goodreau SM, Carnegie NB, Vittinghoff E, et al. What drives the US and Peruvian HIV epidemics in men who have sex with men (MSM)? *PloS one.* 2012;7(11):e50522.
- 29. Mitchell JW, Petroll AE. HIV testing rates and factors associated with recetn HIV testing among male couples. *Sexually Transmitted Diseases*. 2012;39(5):379-381.
- 30. Stephenson R, White D, Darbes L, Hoff CC, Sullivan P. HIV testing behaviors and perceptions of risk of HIV infection among MSM with main partners. *AIDS Behav.* 2015;19:553-560.
- 31. Starks TJ, Golub SA, Payton G, Weinberger C, Parsons JT. Contextualizing condom use: Stigma, intimacy interfearance, and unprotected sex. *J Health Psychol.* 2014;19(6):711-720.
- 32. Golub SA, Starks TJ, Payton G, Parsons JT. The critical role of intimacy in the sexual risk behaviors of gay and bisexual men. *AIDS Behav.* 2012;16(3):626-632.
- 33. Mutchler MG. Young gay men's stories in the states: Scripts, sex, and safty in the time of AIDS. *Sexualities*. 2000;3(1):31-54.
- 34. Campbell CK, Gomez AM, Dworkin S, et al. Health, trust, or "Just Understood": explicit and implicit condom decisionmaking processes among black, white, and interracial same-sex male couples. *Archives of Sexual Behavior*. 2014;43:697-706.



- 35. Mustanski B, Newcomb ME, Clerkin EM. Relationship characteristics and sexual risk-taking in young men who have sex with men. *Health Psychology*. 2011.
- 36. Starks TJ, Grov C, Parsons JT. Sexual compulsivity and interpersonal functioning: sexual relationship quality and sexual health in gay relationships. *Health Psychol*. 2013;32(10):1047-1056.
- 37. Rusbult CE, Bissonnette VL, Arriaga XB, Cox CL, Bradbury TN. Accommodation processes during the early years of marriage. *The developmental course of marital dysfunction*. 1998:74-113.
- 38. Rusbult CE, Verette J, Whitney GA, Slovik LF, Lipkus I. Accommodation processes in close relationships: Theory and preliminary empirical evidence. *Journal of Personality and Social Psychology.* 1991;60(1):53-78.
- 39. Yovetich NA, Rusbult CE. Accommodative behavior in close relationships: Exploring transformation of motivation. *Journal of Experimental Social Psychology*. 1994;30(2):138-164.
- 40. Lewis MA, Gladstone E, Schmal S, Darbes LA. Health-related social control and relationship interdependence among gay couples. *Health Education Research*. 2006;21(4):488-500.
- 41. Hoff CC, Beougher SC, Chakravarty D, Darbes LA, Neilands TB. Relationship characteristics and motivations behind agreements among gay male couples:

  Differences by agreement type and couple serostatus. *AIDS Care*. 2010;22(7):827-835.
- 42. Parsons JT, Starks TJ, DuBois S, Grov C, Golub SA. Alternatives to monogamy among gay male couples in a community survey: Implications for mental health and sexual risk. *Arch Sex Behav.* 2013;42(2):303-312.
- 43. Parsons JT, Starks TJ, Gamarel KE, Grov C. (Non)monogamy and sexual relationship quality among same-sex male couples. *Journal of Family Psychology*. 2012;26(5):669-677.
- 44. Grov C, Starks TJ, Rendina HJ, Parsons JT. Rules about casual sex partners, relationship satisfaction, and HIV risk in partnered gay and bisexual men. *Journal of Sex and Marital Therapy.* 2014;40(2):105-122.
- 45. Parsons JT, Starks TJ, Grov C. Understanding the role of sexual compulsivity and arrangement on the quality of same-sex relationships: An application of the actorpartner model. Annual Meeting of the Society for the Scientific Study of Sexuality; 2011; Houston, TX.
- 46. Starks TJ, Gamarel KE, Johnson MO. Relationship characteristics and HIV transmission risk in same-sex male couples in HIV sero-discordant relationships. *Archives of Sexual Behavior*. 2014;43(1):139-147.
- 47. Gay and Bisexual Men's Health: Substance Abuse. 2013. http://www.cdc.gov/msmhealth/substance-abuse.htm.
- 48. Lanfear C, Akins S, Mosher C. Examining the relationship of substance use and sexual orientation. *Deviant Behavior*. 2013;34(7):586-597.
- 49. Bolton SL, Sareen J. Sexual orientation and its relation to mental disorders and suicide attempts: Findings from a nationally representative sample. *The Canadian Journal of Psychiatry / La Revue canadienne de psychiatrie*. 2011;56(1):35-43.



- 50. Corliss HL, Rosario M, Wypij D, Wylie SA, Frazier AL, Austin SB. Sexual orientation and drug use in a longitudinal cohort study of US adolescents. *Addictive behaviors*. 2010;35(5):517-521.
- 51. Parsons JT, Grov C, Kelly BC. Club drug use and dependence among young adults recruited through time-space sampling. *Public Health Reports*. 2009;124(2):246-254.
- 52. McCabe SE, Boyd C, Hughes TL, d'Arcy H. Sexual identity and substance use among undergraduate students. *Substance Abuse*. 2003;24(2):77-91.
- 53. Schulenberg JE, Magg JL, Steinman KJ, Zucker RA. Development matters: Taking the long view on substance use etiology and intervention during adolescence. In: Monti PM, Colby SM, O'Leary TA, eds. *Adolescents, alcohol, and substance abuse: Reachign teens through brief interventions*. New York: Guilford Press; 2001:19-57.
- 54. Arnett JJ. Emerging adulthood: A theory of development from the late teens through the twenties. *American Psychologist*. 2000;55(5):469-480.
- 55. Newcomb ME, Ryan DT, Greene GJ, Garofalo R, Mustanski B. Prevalence and patterns of smoking, alcohol use, and illicit drug use in young men who have sex with men. *Drug Alcohol Depend*. 2014;141:65-71.
- 56. Mitchell JW, Boyd C, McCabe S, Stephenson R. A cause for concern: Male couples' sexual agreements and their use of substances with sex. *AIDS Behav.* 2014;18(7):1401-1411.
- 57. Grant RM, Lama JR, Anderson PL, et al. Preexposure Chemoprophylaxis for HIV Prevention in Men Who Have Sex with Men. *New England Journal of Medicine*. 2010;363(27):2587-2599.
- 58. USFDA. FDA approves first medication to reduce HIV risk. 2012; http://www.fda.gov/forconsumers/consumerupdates/ucm311821.htm. Accessed April 3, 2015.
- 59. Volk JE, Marcus JL, Phengrasamy T, et al. No new HIV infections with increasing use of HIV preexposure prophylaxis in a clinical practice setting. *Clinical infectious diseases : an official publication of the Infectious Diseases Society of America*. 2015;61(10):1601-1603.
- 60. Liu AY, Cohen SE, Vittinghoff E, et al. Preexposure Prophylaxis for HIV Infection Integrated With Municipal- and Community-Based Sexual Health Services. *JAMA Intern Med.* 2016;176(1):75-84.
- 61. Marrazzo J, Ramjee G, Nair G, et al. Pre-exposure prophylaxis for HIV in women: daily oral tenofovir, oral tenofovir/emtricitabine, or vaginal tenofovir gel in the VOICE study (MTN 003). 20th Conference on Retroviruses and Opportunistic infections GA: Atlanta.
- 62. Van Damme L, Corneli A, Ahmed K, et al. Preexposure prophylaxis for HIV infection among African women. *New England Journal of Medicine*. 2012;367(5):411-422.
- 63. Muganzi D, Boum Y, Musinguzi N, al. e. Comparison of adherence measures in a clinical trial of preexposure prophylaxis. . 2016, February; Seattle, Washington
- 64. Gandhi M, Glidden DV, Liu A, et al. Concentrations of TFV-DP/FTC-TP in dried blood spots and TFV/FTC in hair are strongly correlated in iPrEx OLE. *Journal of Infectious Diseases*. 2015;212(9):1402-1406.
- 65. US Public Health Service. Preexposure prophylaxis for the prevention of HIV infection in the United States—2014: a clinical practice guideline. *Washington, DC: US Public Health Service*. 2014.



- 66. Mitchell JW, Stephenson R. HIV-Negative Partnered Men's Willingness to Use Pre-Exposure Prophylaxis and Associated Factors Among an Internet Sample of U.S. HIV-Negative and HIV-Discordant Male Couples. *LGBT Health*. 2015;2(1):35-40.
- 67. Solomon MM, Mayer KH, Glidden DV, et al. Syphilis predicts HIV incidence among men and transgender women who have sex with men in a preexposure prophylaxis trial. *Clinical Infectious Diseases*. 2014;59(7):1020-1026.
- 68. Parsons JT, Rendina HJ, Lassiter JM, Whitfield THF, Starks TJ, Grov C. Uptake of HIV preexposure prophylaxis (PrEP) in a national sample of gay and bisexual men in the United States: The Motivational PrEP Cascade. *Journal of Acquired Immune Deficiency Syndrome*. in press.
- 69. Holloway IW, Dougherty R, Gildner J, et al. Brief Report: PrEP uptake, adherence, and discontinuation among Calivornia YMSM using geosocial netowkring applications. Journal of Acquired Immune Deficiency Syndrome. 2017;74(1):15-20.
- 70. Gamarel KE, Golub SA. Intimacy motivations and pre-exposure prophylaxis (PrEP) adoption intentions among HIV-negative men who have sex with men (MSM) in romantic relationships. *Annals of Behavioral Medicine*. 2015;49(2):177 186.
- 71. Gamarel KE, Golub SA. Intimacy motivations and pre-exposure prophylaxis (PrEP) adoption intentions among HIV-negative men who have sex with men (MSM) in romantic relationships. *Ann Behav Med.* 2015;49(2):177 186.
- 72. Rendina HJ, Whitfield THF, Grov CS, T.J., Parsons JT. Distinguishing hypothetical willingness from behavioral intentions to initiate HIV pre-exposure prophylaxis (PrEP): Findings from a large cohort of gay and bisexual men in the U.S. *Social Science & Medicine*. in press.
- 73. Mimiaga MJ, Closson EF, Kothary V, Mitty JA. Sexual partnerships and considerations for HIV antiretroviral pre-exposure prophylaxis utilization among high-risk substance using men who have sex with men. *Arch Sex Behav.* 2014;43(1):99-106.
- 74. Miller WR, Rollnick S. *Motivational Interviewing*. 3rd ed. New York: Guilford Press; 2013.
- 75. Miller WR, & Rollnick, S. P. *Motivational Interviewing, Third Edition: Helping People Change* Guilford Press; 2012.
- 76. D'Amico EJ, Miles JNV, Stern SA, Meredith LS. Brief motivational interviewing for teens at risk of substance use consequences: A randomized pilot study in a primary care clinic. *Journal of Substance Abuse Treatment*. 2008;35(1):53-61.
- 77. Naar-King S, Parsons JT, Murphy DA, Kolmodin K, Harris DR. A multisite randomized trial of a motivational intervention targeting multiple risks in youth living with HIV: Initial effects on motivation, self-efficacy, and depression. *Journal of Adolescent Health*. 2010;46(5):422-428.
- 78. Naar-King S, Wright K, Parsons JT, et al. Health Choices: Motivational enhancement therapy for health risk behaviros in HIV-positive youth. *AIDS Education & Prevention*. 2006;18(1):1-11.
- 79. Stephenson R, Rentsch C, Sullivan PS. High levels of acceptability of couples-based HIV testing among MSM in South Africa. *AIDS Care*. 2012;24(4):529-535.
- 80. Fals-Stewart W, O'Farrell TJ, Lam WKK. Behavioral couples therapy for gay and lesbian couples with alcohol use disorders. *Journal of Substance Abuse Treatment*. 2009;37(4):379-387.



- 81. Erikson EH. *Identity: Youth and crisis.* New York: Norton; 1968.
- 82. Rew LW, Taylor-Seehafer TA, Smith MA, Lorie R. Sexual health risks and protective resources in gay, lesbian, bisexual, and heterosexual homeless youth. *Journal of Specialists in Pediatric Nursing*. 2005;10(1):11-19.
- 83. Remafedi G. Predictors of unprotected intercourse, amogn gay and bisexual youth: Knowledge, beliefs, and behavior. *Pediatrics*. 1994;94(2):163-168.
- 84. Rotheram-Borus MJ, Reid H, Rosario M, Kasen S. Determinants of safer sex patters among gay/bisexual male adolescents. *Journal of Adolescence*. 1995;18:3-15.
- 85. United States Drug Testing Laboratories I. Fingernail drug testing. 2016; http://www.usdtl.com/testing/fingernail-drug-test-labs. Accessed 5/5/2016, 2016.
- 86. Starks TJ, Payton G, Golub SA, Weinberger C, Parsons JT. Contextualizing condom use: Intimacy interference, stigma, and unprotected sex. *J Health Psychol.* 2014;19(6):711-720.
- 87. Starks TJ, Millar BM, Tuck A, Wells B. The role of sexual expectancies of substance use as a mediator between adult attachment and drug use among gay and bisexual men. *Drug Alcohol Depend*. 2015.
- 88. Starks TJ, Parsons JT. Adult attachment among partnered gay men: Patterns and associations with sexual relationship quality. *Archives of Sexual Behavior*. 2014;43(1):107-117.
- 89. Gamarel KE, Starks TJ, Dillworth SE, Neilands T, Taylor JM, Johnson MO. Personal or relational? Examining sexual health in the context of HIV serodiscordant same-sex male couples. *AIDS Behav.* 2014;18(171-179).
- 90. Starks TJ, Tuck A, Millar BM, Parsons JT. Linking syndemic stress and behavioral indicators of HIV transmission risk in gay couples. *AIDS Behav.* 2016;20(2):439-448.
- 91. Starks TJ, Castro MA, Miller BM, Castiblanco JP. Modeling interpersonal correlates of condomless anal sex among gay and bisexual men: An application of attachment theory. under review.
- 92. Moyers TB, Martin T, Manuel JK, Hendrickson SML, Miller WR. Assessing competence in the use of motivational interviewing. *J Subst Abuse Treat*. 2005;28(1):19-26.
- 93. Murphy DA, Chen X, Naar-King S, Parsons JT. Alcohol and marijuana use outcomes in the Healthy Choices Motivational Interviewing Intervention for HIV-positive youth. *AIDS Patient Care and STDs.* 2012;26 (2):95-100.
- 94. Miller PM, Anton RF. Biochemical alcohol screening in primary health care. *Addictive Behaviors*. 2004;29:1427-1437.
- 95. Williams AB, Rivet Amico K, Bova C, Womack JA. A proposal for quality standards for measuring medication adherence in research. *AIDS & Behavior*. 2012;Epub ahead of print.
- 96. Kelley C, Kahle E, Siegler A, et al. Applying a PrEP continuum of care for men who have sex with men in Atlanta, Georgia. *Clin Infect Dis.* 2015;61(10):1590 1597.
- 97. Prochaska JO, Velicer WF. The transtheoretical model of health behavior change. *Am J Health Promot.* 1997;12(1):38-48.
- 98. Velicer WF, Prochaska JO, Fava JL, Norman GJ, Redding CA. Smoking cessation and stress management: Applications of the transtheoretical model of behavior change. *Homeost Health Dis.* 1998;38(5):216-233.



- 99. Sullivan PS, White D, Rosenberg ES, et al. Safety and acceptability of couples HIV testing and counseling for US men who have sex with men: a randomized prevention study.

  Journal of the International Association of Physicians in AIDS Care. 2014;13(2):135-144.
- 100. Neilands TB, Chakravarty D, Darbes LA, Beougher SC, Hoff CC. Development and validation of the sexual agreement investment scale. *The Journal of Sex Research*. 2009;47(1):24-37.
- 101. Hoff CC, Chakravarty D, Beougher SC, Darbes LA, Dadasovich R, Neilands TB. Serostatus differences and agreements about sex with outside partners among gay male couples. *AIDS Education & Prevention*. 2009;21(1):25-38.
- 102. Mustanski B, Newcomb ME, Clerkin EM. Relationship characteristics and sexual risk-taking in young men who have sex with men. *Health Psychol.* 2011;30(5):597-605.
- 103. First MB, Gibbon M, Spitzer R, Williams J. User's guide for the Structured Clinical Interview for DSM-IV Axis I Disorders Research version SCID-I, Version 2. 1996.
- 104. Folstein MF, Folstein SE, McHugh RR. Mini-mental state: A practical method for grading the cognitive state of patients for the clinician. *Journal of Psychiatric Research*. 1975;12:189-198.
- 105. Parsons JT, Vial AC, Starks TJ, Golub SA. Recruiting drug-using men who have sex with men in behavioral intervention trials: A comparison of internet-based and field-based strategies. *AIDS Behav.* 2013;17(2):688-699.
- 106. Vial AC, Starks TJ, Parsons JT. Finding and recruiting the highest risk HIV-negative men who have sex with men. *AIDS Education & Prevention*. 2014;26(1):56-67.
- 107. NHBS. National HIV Behavioral Surveillance System: Heterosexuals at Increased Risk of HIV. 2010:1-352.
- 108. Skinner HA. The drug abuse screening test. *Addict Behav.* 1982;7(4):363-371.
- 109. Carey MP, Schroder KE. Development and psychometric evaluation of the brief HIV Knowledge Questionnaire. *AIDS education and prevention: official publication of the International Society for AIDS Education*. 2002;14(2):172-182.
- 110. Prochaska JO, Velicer WF, Rossi JS, et al. Stages of change and decisional balance for 12 problem behaviors. *Health Psychol.* 1994;13(1):39-46.
- 111. Annis HM, Martin G. *Drug-taking confidence questionnair*. Toronto, Canada: Addiction Research Foundation. Centre for Addiction and Mental Health; 1985.
- 112. Forsyth AD, Carey MP, Fuqua RW. Evaluation of the validity of the Condom Use Self-Efficacy Scale (CUSES) in young men using two behavioral simulations. *Health Psychol*. 1997;16(2):175.
- 113. Johnson MO, Neilands TB, Dilworth SE, Morin SF, Remien RH, Chesney MA. The role of self-efficacy in HIV treatment adherence: validation of the HIV Treatment Adherence Self-Efficacy Scale (HIV-ASES). *J Behav Med.* 2007;30(5):359-370.
- 114. Derogatis LR, Melisaratos N. The brief symptom inventory: an introductory report. *Psychological Medicine*. 1983;13(3):595-605.
- 115. Stucky BD, Gottfredson NC, Panter AT, Daye CE, Allen WR, Wightman LF. An item factor analysis and item response theory-based revision of the everyday discrimination scale. *Cultural Diversity and Ethnic Minority Psychology.* 2011;17(2):175-185.
- 116. Stephenson R, Finneran C. The IPV-GBM scale: a new scale to measure intimate partner violence among gay and bisexual men. *PLoS ONE*. 2013;8(6):e62592.



- 117. Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. *Addiction*. 1993;88(6):791-804.
- 118. Busby DM, Christensen C, Crane DR, Larson JH. A revision of the dyadic adjustment scale for use with destressed and nondistressed couples: Construct hierarchy and multidimensional scales. *Journal of Marital and Family Therapy.* 1995;21(3):289-308.
- 119. Rubin RB, Martin MM. Development of a measure of interpersonal competence. *Communication Research Reports.* 1994;11(1):33-44.
- 120. Christensen C, Shenk JL. Communication, conflict, and psychological distance in nondistressed, clinic, and divorcing couples. *Journal of Consulting and Clinical Psychology.* 1991;59(458-463).
- 121. Catania JA. Dyadic sexual communication scale. In: Davis CM, Yarber WL, Bauserman R, Schreer G, Davis SL, eds. *Handbook of sexuality-related measures*. Thousand Oaks, CA: SAGE Publications, Inc.; 1998:129-130.
- 122. Salazar LF, Stephenson RB, Sullivan PS, Tarver R. Development and validation of HIV-related dyadic measures for men who have sex with men. *Journal of Sex Research*. 2013;50(2):164-177.
- 123. Lehmiller JJ, Agnew CR. Marginalized relationships: The impact of social disapproval on romantic relationship commitment. *Personality and Social Psychology Bulletin*. 2006;32(1):40-51.
- 124. Pulerwitz J, Gortmaker SL, DeJong W. Measuring sexual relationship power in HIV/STD research. *Sex Roles*. 2000;42(7/8):637-660.
- 125. Sobell LC, Sobell MB. *Timeline followback user's guide.* Toronto: Alcohol Research Foundation; 1996.
- 126. Sobell MB, Sobell LC. *Problem drinkers: Guided self-change treatment.* New York: Guilford Press; 1993.
- 127. Carey KB, Maisto SA, Carey MP, Purnine DM. Measuring readiness-to-change substance misuse among psychiatric outpatients: I. Reliability and validity of self-report measures. *J Stud Alcohol.* 2001;62(1):79-88.
- 128. Weinhardt LS, Carey MP, Maisto SA, Carey KB, Cohen MM, Wickramasinghe SM. Reliability of the timeline follow-back sexual behavior interview. *Ann Behav Med.* 1998;20(1):25-30.
- 129. Fals-Stewart W, O'Farrell TJ, Freitas TT, McFarlin SK, Rutigliano P. The timeline followback reports of psychoactive substance use by drug-abusing patients: psychometric properties. *Journal of Consulting and Clinical Psychology.* 2000;68(1):134-144.
- 130. R.M. G, P.L. A, V. M, et al. Uptake of pre-exposure prophylaxis, sexual practices, and HIV incidence in men and trnasgender women who have sex with men: A cohort study. *The Lancet*. 2014;14(9):820-829.
- 131. J.R. C-M, H. ZJ, J.E. R, et al. Tenofovir, emtricitabine, and tenofovir diphosphate in dried blood spots for determining recent and cumulative drug exposure. *AIDS Research and Human Retroviruses*. 2013;29(2):384-390.



- 132. DiFrancesco R, Tooley K, Rosenkranz SL, et al. Clinical Pharmacological Therapy. *2013*. Clinical pharmacology quality assurance for HIV and related infectious diseases research;93(6):479-482.
- 133. Del Boca FK, Noll JA. Truth or consequences: the validity of self-report data in health services research on addictions. *Addiction*. 2000;95(11s3):347-360.
- 134. Dowling-Guyer S, M.E. J, D.G. F, al. e. Reliability of drug users' self-reported HIV risk behaviors and validity of self-reported recent drug use. *Assessment*. 1994;1(4):383-392.
- 135. Harrison LD, Martin SS, Enev T, Harrington D. *Comparing drug testing and self-report of drug use among youths and young adults in the general population.* Department of Health and Human Services, Substance Abuse and Mental Health Services Administration, Office of Applied Studies; 2007.
- 136. Williams ML, Freeman RC, Bowen AM, Z Z. A comparison of the reliability of self-reported drug use and sexual behaviors using computer-assisted versus face-to-face interviewing. *AIDS Education & Prevention*. 2000;12(3):199.
- 137. Babor TF, Brown J, del Boca FK. Validity of self-reports in applied research on addictive behaviors: Fact or fiction? *Behavioral Assessment*. 1990.
- 138. Identigene. Identigene STD Test Collection Kit. 2011; http://www.identigene.com/std-testing/.
- 139. Gene-Probe. APTIMA COMBO 2® Assay. 2011; http://www.gen-probe.com/products-services/aptima.aspx.
- 140. Kratz M, Terranova E, Fuld J. Provider reporting: How to report diseases, events, and conditions to the New York City Health Department. New York, NY: The New York City Department of Health and Mental Hygiene; 2015.
- 141. Moyers TB, Manuel JK, Ernst D. *Motivational Interviewing Treatment INtegrity Coding Manual 4.0.* Unpublished manual; 2014.
- 142. NCSS, Hintze JL. PASS: Power Analysis and Sample Size System. Kaysville, Utah2011.
- 143. Starks TJ. Condom use in gay couples: examining communication and identifying motivations. Conference on contemporary issues in Gay Men's Sexual Health Research; April, 2016, 2016; Puerto Vallarta.
- 144. Patton M. *Qualitative research and evaluation methods.* 3rd ed. Thousand Oaks, CA: Sage; 2000.
- 145. Goodenough W. Describing a Culture. *Description and Comparison in Cultural Anthropology*: Cambridge University Press; 1970:104 119.
- 146. Vial AC, Starks TJ, Parsons JT. Relative efficiency of field and online strategies in the recruitment of HIV-positive men who have sex with men. *AIDS Educ Prev*. 2015;27(2):103-111.